CLINICAL TRIAL: NCT00192452
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study of MEDI-507, a Humanized Monoclonal Antibody That Binds to the CD2 Receptor, Administered by Intravenous Infusion to Adults With Plaque Psoriasis
Brief Title: Study of MEDI-507 Administered by Intravenous Infusion to Adults With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP074
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2006-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — siplizumab

INTERVENTIONS:
Drug: MEDI-507

SUMMARY:
- The primary objective of this study is to compare disease activity, as measured by PASI score, of two MEDI-507 dose levels (0.012 and 0.04 mg/kg) versus placebo administered by intravenous infusion every 2 weeks for a total of 8 infusions.

ELIGIBILITY:
Inclusion Criteria:

* Plaque psoriasis involving at least 10% of body surface area (Appendix B)
* Age 18 through 65 years at the time of the first dose of study drug
* Both males and females are eligible. However, sexually active females, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 30 days prior to the first dose of study drug and must agree to continue using such precautions for 60 days after the final dose of study drug
* Currently receiving no therapy for psoriasis except emollients (certain other over-the-counter products may be allowed with prior approval of the sponsor)
* Written informed consent obtained from the patient
* Ability to complete follow-up period of 188 days as required by the protocol

Exclusion Criteria:

* Pustular, guttate, or erythrodermic psoriasis as the predominant disease type
* PASI score <8
* At screening (must be within 21 days before study entry) any of the following: lymphocyte count under 1,200 cells/mm3, WBC under 4,000 cells/mm3, hematocrit below 32%, platelets below 110,000 cells/mm3, creatinine, AST, ALT over 1.5 times upper limit of normal
* At screening (must be within 21 days before study entry) any clinical evidence of HIV, hepatitis B, hepatitis C or active hepatitis A infection
* Pregnancy (must have a negative serum pregnancy test within 21 days prior to the first dose of study drug, and urine pregnancy test must be negative on Study Day 0 before study entry)
* History of cancer (except excision of basal cell carcinoma)
* Any documented immunodeficiency
* A history of prior administration of monoclonal antibodies or related proteins, with the exception of MEDI-507 (Note: prior recipients of MEDI-507 will require review and approval by the sponsor prior to entry)
* Receipt of systemic retinoids, corticosteroids, cyclosporin A, methotrexate, phototherapy or coal tar treatment in the past 4 weeks
* Use of topical therapy (except emollients) for psoriasis in the past 2 weeks (certain other over-the-counter products may be allowed with prior approval of the sponsor)
* Receipt of any investigational drug therapy within 6 weeks before the first dose of study drug in this protocol (use of licensed agents for indications not listed in the package insert is permitted)
* Current or planned participation in a research protocol in which an investigational agent or therapy may be administered
* Nursing mother
* Acute illness including infections
* Clinical manifestations of significant end organ dysfunction or failure that may compromise the safety of the volunteer in the study
* A known drug allergy or medical contraindication to ibuprofen

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2001-03; Study Completion 2001-12

PRIMARY OUTCOMES:
Analyses of categorical data will be performed and analysis of continuous data will be performed using a one-way analysis of variance (ANOVA) with traetment group as a factor.

SECONDARY OUTCOMES:
Percentage of subjects with at least 75% improvement and those with at least 50% improvement will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Pillemer, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - MDS Pharma Services (US) Inc., Phoenix, Arizona
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Northwest Kinetics, Tacoma, Washington